CLINICAL TRIAL: NCT03278964
Title: Comparative Morphometric, Functional and Psychosocial Analysis Between the Results of Two Surgical Techniques of Orbital Decompression in Patients With Graves Orbitopathy
Brief Title: Analysis Between the Results of Two Surgical Techniques of Orbital Decompression in Patients With Graves Orbitopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Cristiane de Almeida Leite, Medical Doctor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 39748114.0.0000.0068
Record Dates: First submitted 2017-09-04; First posted 2017-09-12 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Graves Ophthalmopathy
Keywords: Graves Disease; Orbital decompression; Graves Orbitopathy; Exophthalmos; Diplopia; Restrictive Strabismus
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease; Exophthalmos; Diplopia

STUDY DESIGN:
Intervention Model Description: Patients with Graves orbitopathy will be randomly divided in two groups. One group will be submmited to orbital decompression by antro-ethmoidal technique. The other group will be treated by lateral wall technique.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and investigators do not know which orbital decompression technique will be done until 6 months of postoperative period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antro-ethmoidal technique (Active Comparator): Patients in the inactive phase of Graves orbitopathy will be submitted to orbital decompression by antro-ethmoidal technique.
  Interventions: Procedure: Orbital decompression
- Lateral wall technique (Experimental): Patients in the inactive phase of Graves orbitopathy will be submitted to orbital decompression by lateral wall technique.
  Interventions: Procedure: Orbital decompression

INTERVENTIONS:
Procedure: Orbital decompression

SUMMARY:
Randomized prospective clinical trial, aiming to compare two techniques of orbital decompression. Patients with Graves orbitopathy in the inactive phase for at least 6 months will be divided in two groups; one group will be submitted to orbital decompression by antro-ethmoidal technique; the other group will be submitted to orbital decompression by lateral wall technique. Patients will be followed up for a period of 6 months after the surgery, and will be evaluated about the effect of orbital decompression on ocular motility, proptosis, ocular surface and quality of life.

DETAILED DESCRIPTION:
Graves' orbitopathy is the most relevant non-thyroid manifestation of Graves' disease. Its clinical status varies from subclinical to severe deformities. Clinical features include palpebral retraction, exophthalmos, restrictive strabismus, chemosis, ocular surface lesions and optic neuropathy. There are two stages of the disease. There is an active phase in which the inflammatory process is present and the orbital changes evolve. The inactive phase comprises a stable clinical picture regarding the sequelae of the active phase. Orbital decompression surgery is the main treatment procedure for this inactive phase for functional and cosmetic rehabilitation purposes. In the last decades, great advances in the techniques and indication of this surgery have been observed. However, a consensus about the ideal technique does not yet exist. The most commonly used techniques are antro-ethmoidal decompression and lateral wall decompression alone or associated with other walls. The present study will be based on patients with Graves' orbitopathy diagnosis for at least 2 years and who are already in the inactive phase for at least 6 months. There are no prospective studies comparing the 2 main orbital decompression techniques through a detailed analysis of surgical outcomes from computed tomography images, digital photographic images and ocular motility examination. These informations will be collected in the preoperative and postoperative periods. The investigators will evaluate the decompressive potential of each technique calculated by the tomographic images. Participants will be followed up for a period of 6 months after the surgical procedure and the effect of decompression on ocular motility, ocular bulb positioning, ocular surface, vertical palpebral fissure, and the patient's quality of life will also be analyzed. The findings of this work will bring important contribution to the improvement of this surgical procedure of great relevance in the rehabilitation of patients with Graves' orbitopathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Graves orbitopathy for at least 2 years
* Clinical Activity Score (CAS) < 4 for at least 6 months
* Agreement with the Informed Consent Form, which will be signed during the selection visit
* Ability to come to periodic evaluations for 6 months after the orbital decompression
* Absence of ocular abnormalities such as degenerative myopia, microphthalmia or anophthalmic cavity
* Absence of orbital abnormalities such as previous fractures or congenital defects
* Good collaboration for the exams
* Euthyroidism
* Exophthalmus ≥ 20 mm in Hertel's exophthalmometry
* Preoperative clinical evaluation indicating absence of contraindications for a surgical procedure

Exclusion Criteria:

* Myasthenia gravis
* Pregnancy
* Previous orbital, strabismus or eyelid surgery
* Other abnormal eye conditions or symptoms that make it impossible to admit the patient to the study, according to the clinical judgment of the investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Ocular Motility status | Before orbital decompression and 1, 3 and 6 months after surgery
  Measure by prism and cover, to assess strabismus in the nine positions of gaze
Exophthalmos | Before orbital decompression and 6 months after surgery
  Exophthalmos will be measured by Hertel's exophthalmometer and orbital computerized tomography

SECONDARY OUTCOMES:
Diplopia | Before orbital decompression and 1, 3 and 6 months after surgery
  Evaluation by Gorman's Diplopia Table
Digital photography evaluation | Before orbital decompression and 6 months after surgery
  Using digital photography, Photoshop and Image J, ductions and versions will be analyzed
Volume of the extraocular muscles | Before orbital decompression and 6 months after surgery
  Measure by orbital computerized tomography images
Ocular surface evaluation | Before orbital decompression and 6 months after surgery
  Assessed by Lysozyme Green, Break-up time, Schirmer I test
Quality of life questionary Quality of life questionary | Before orbital decompression and 6 months after surgery
  GO-QoL form

CONTACTS AND LOCATIONS:
Overall Officials: MARIO L RIBEIRO MONTEIRO, PHD, Study Chair — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leite CA, Pereira TS, Chiang J, Moritz RB, Goncalves ACP, Monteiro MLR. Ocular motility changes after inferomedial wall and balanced medial plus lateral wall orbital decompression in Graves' orbitopathy: a randomized prospective comparative study. Clinics (Sao Paulo). 2021 Apr 9;76:e2592. doi: 10.6061/clinics/2021/e2592. eCollection 2021. PMID 33852655
- [Derived] Leite CA, Pereira TS, Chiang J, Pieroni Goncalves AC, Monteiro MLR. Evaluation of Ocular Versions in Graves' Orbitopathy: Correlation between the Qualitative Clinical Method and the Quantitative Photographic Method. J Ophthalmol. 2020 Jul 31;2020:9758153. doi: 10.1155/2020/9758153. eCollection 2020. PMID 32832143